CLINICAL TRIAL: NCT02801747
Title: Using MOST to Optimize an HIV Care Continuum Intervention for Vulnerable Populations
Acronym: HTH2-MOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Penn State University (Other); Binghamton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: i15-01480
Record Dates: First submitted 2016-06-08; First posted 2016-06-16 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-07

CONDITIONS: HIV
Keywords: HIV care continuum; antiretroviral therapy; engagement in HIV care; Multiphase Optimization Strategy (MOST)

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Condition 1 (Experimental): Receives a core intervention session and the navigation intervention component (long duration; that is, up to 6 months).
  Interventions: Behavioral: Heart to Heart2 (HTH2)
- Condition 2 (Experimental): Receives a core intervention session, the focused support group component, and the navigation intervention component (short duration, that is, up to 3 months).
  Interventions: Behavioral: Heart to Heart2 (HTH2)
- Condition 3 (Experimental): Receives a core intervention session, the peer mentorship component, and the navigation intervention component (short duration, that is, up to 3 months).
  Interventions: Behavioral: Heart to Heart2 (HTH2)
- Condition 4 (Experimental): Receives a core intervention session, the peer mentorship component, the focused support group component, and the navigation intervention component (long duration, that is, up to 6 months).
  Interventions: Behavioral: Heart to Heart2 (HTH2)
- Condition 5 (Experimental): Receives a core intervention session, the pre-adherence preparation component, and the navigation intervention component (short duration, that is, up to 3 months).
  Interventions: Behavioral: Heart to Heart2 (HTH2)
- Condition 6 (Experimental): Receives a core intervention session, the pre-adherence preparation component, the focused support group component, and the navigation intervention component (long duration, that is, up to 6 months).
  Interventions: Behavioral: Heart to Heart2 (HTH2)
- Condition 7 (Experimental): Receives a core intervention session, the pre-adherence preparation component, the peer mentorship component, and the navigation intervention component (long duration, that is, up to 6 months).
  Interventions: Behavioral: Heart to Heart2 (HTH2)
- Condition 8 (Experimental): Receives a core intervention session, the pre-adherence preparation component, the peer mentorship component, and the navigation intervention component (short duration, that is, up to 3 months).
  Interventions: Behavioral: Heart to Heart2 (HTH2)
- Condition 9 (Experimental): Receives a core intervention session, the Motivational Interviewing sessions component, and the navigation intervention component (short duration, that is, up to 3 months).
  Interventions: Behavioral: Heart to Heart2 (HTH2)
- Condition 10 (Experimental): Receives a core intervention session, the Motivational Interviewing sessions component, the focused support group component, and the navigation intervention component (long duration, that is, up to 6 months).
  Interventions: Behavioral: Heart to Heart2 (HTH2)
- Condition 11 (Experimental): Receives a core intervention session, the Motivational Interviewing sessions component, the peer mentorship component, and the navigation intervention component (long duration, that is, up to 6 months).
  Interventions: Behavioral: Heart to Heart2 (HTH2)
- Condition 12 (Experimental): Receives a core intervention session, the Motivational Interviewing sessions component, the peer mentorship component, the focused support group component, and the navigation intervention component (short duration, that is, up to 3 months).
  Interventions: Behavioral: Heart to Heart2 (HTH2)
- Condition 13 (Experimental): Receives a core intervention session, the Motivational Interviewing sessions component, the pre-adherence preparation component, and the navigation intervention component (long duration, that is, up to 6 months).
  Interventions: Behavioral: Heart to Heart2 (HTH2)
- Condition 14 (Experimental): Receives a core intervention session, the Motivational Interviewing sessions component, the pre-adherence preparation component, the focused support group component, and the navigation intervention component (short duration, that is, up to 3 months).
  Interventions: Behavioral: Heart to Heart2 (HTH2)
- Condition 15 (Experimental): Receives a core intervention session, the Motivational Interviewing sessions component, the pre-adherence preparation component, the peer mentorship component, and the navigation intervention component (short duration, that is, up to 3 months).
  Interventions: Behavioral: Heart to Heart2 (HTH2)
- Condition 16 (Experimental): Receives a core intervention session, the Motivational Interviewing sessions component, the pre-adherence preparation component, the peer mentorship component, the focused support group component, and the navigation intervention component (long duration, that is, up to 6 months).
  Interventions: Behavioral: Heart to Heart2 (HTH2)

INTERVENTIONS:
Behavioral: Heart to Heart2 (HTH2) — The present study uses a fractional factorial design to evaluate the efficacy of five distinct culturally appropriate intervention components on the primary outcome, HIV viral suppression.

SUMMARY:
The present study targets the large population of persons living with HIV/AIDS (PLHA) in the U.S. who are both insufficiently engaged in HIV primary care and not taking antiretroviral therapy (ART), who are mainly African American/Black and Latino. NIH has emphasized the urgent need for new research approaches to advance intervention science, and the proposed project employs a new, potent, and innovative research methodology, the Multiphase Optimization STrategy (MOST), a framework for developing highly efficacious, efficient, scalable, and cost-effective interventions. The proposed study has the highest public health significance: it addresses a vulnerable population of PLHA, including the critically important subpopulations of men who have sex with men (MSM) and substance users; will develop an efficient and cost effective intervention to increase engagement along the HIV care continuum for these vulnerable groups; and addresses two areas highlighted in the August 2015 notice on research priorities from the NIH Office of AIDS Research (NOT-OD-15-137), namely, engaging PLHA in prevention/treatment services, and reducing HIV/AIDS-related racial/ethnic disparities.

DETAILED DESCRIPTION:
More than half of persons living with HIV/AIDS (PLHA) in the U.S. are insufficiently engaged in HIV primary care and not taking antiretroviral therapy (ART), mainly African Americans and Latinos. In the proposed project, two experienced and productive behavioral scientists will employ a potent and innovative research methodology, the Multiphase Optimization STrategy (MOST), to develop a highly efficacious, efficient, scalable, and cost-effective intervention to increase engagement along the HIV care continuum. Whereas randomized controlled trials (RCTs) are valuable for evaluating the efficacy of multi-component interventions as a package, they are not designed to evaluate which specific components contribute to efficacy. MOST, a pioneering, engineering-inspired framework, addresses this problem through highly efficient randomized experimentation to assess the performance of individual intervention components and their interactions. The investigators propose to use MOST to engineer an intervention to increase engagement along the HIV care continuum for African American and Latino PLHA not well engaged in care and not taking ART. Further, the intervention will be optimized for cost-effectiveness. This efficiency and cost-effectiveness are critical in a time of constrained resources, and will also increase the intervention's future scalability. NIH has signaled its interest in MOST, and this is the first study to apply it in the field of adult HIV treatment. A similar set of multi-level factors impede both HIV care and ART initiation for African American and Latino PLHA, primary among them individual (e.g., substance use, distrust, fear), social (e.g., stigma), and structural-level barriers (e.g., difficulties accessing ancillary services). Guided by a multi-level social cognitive theory, the study will evaluate 5 distinct intervention components (i.e., Motivational Interviewing sessions, pre-adherence preparation, support groups, peer mentorship, and patient navigation), each designed to address a specific barrier to HIV care and ART initiation. These components are well-grounded in the empirical literature and were found acceptable, feasible, and promising with respect to efficacy in a preliminary study. Study aims are: 1) using a highly efficient experimental design, identify which of 5 components contribute meaningfully to improvement in viral suppression, and secondary outcomes of ART adherence and engagement in HIV primary care; 2) identify mediators and moderators of component efficacy; and 3) using a mathematical modeling approach, build the most cost-effective and efficient intervention package from the efficacious components. A heterogeneous sample of African American and Latino PLHA (with respect to age, substance use, and sexual minority status) will be recruited with a proven hybrid sampling method using targeted sampling in community settings and peer recruitment (N=512). This highly innovative and significant study, which addresses a high-priority research area (NIH NOT-OD-15-137), will produce an HIV care continuum intervention for the nation's most vulnerable PLHA, optimized for cost-effectiveness, and with exceptional levels of efficacy, efficiency, and scalability.

ELIGIBILITY:
Inclusion Criteria:

* African American/Black or Latino/Hispanic race/ethnicity
* HIV diagnosed for at least 6 months (HIV status confirmed with medical documentation)
* Has not taken antiretroviral therapy (ART) in the past 6 weeks (the period of time assessed by hair assay, and a reasonable period of time not on ART for the present study)
* Sub-optimal engagement in HIV care (assessed from the medical record, defined as less than 1 visit in every 4-mo. period in the past year [two of them at least 90 days apart], pro-rated for those diagnosed less than a year ago) or > 2 missed visits (without prior cancellation) in the past year
* Reside in the New York City (NYC) metropolitan area
* Not planning to leave the NYC metropolitan area in next year
* Not actively psychotic based on screening instrument
* Not a participant in the preliminary pilot HTH R34 study
* Able to conduct research activities in English or Spanish
* Willing to provide hair sample (if possible), blood samples (to assess CD4, VL), and Medical Report Form ([MRF]; to assess health care attendance) at screening
* Willing to participate in a Core intervention session and be randomly assigned to 1-5 intervention components.

Exclusion Criteria:

NONE SEE ABOVE

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Change in HIV viral suppression | Assessed at 4 month follow up (FU), 12 month FU
  Blood will be drawn and viral load will be assessed via laboratory report (Bioreference Lab, HIV-1,RNA,PCR,ULTRA). Participants will not have viral suppression at baseline. Change in viral suppression, that is, whether viral suppression has been achieved, will be coded as present if viral load levels are < 20 ppml. Viral suppression will be assessed at both FU periods. Participants may achieve this primary endpoint, or not, at one or both FU periods.

SECONDARY OUTCOMES:
Absolute HIV viral load (log10) | Assessed at baseline, 4 month follow up (FU), 12 month FU
  Blood will be drawn and viral load will be assessed via laboratory report (Bioreference Lab, HIV-1,RNA,PCR,ULTRA).
Adherence to antiretroviral therapy | 4 month follow up (FU), 8 month FU, 12 month FU
  Hair samples will be tested for average adherence to antiretroviral therapy
Engagement in HIV primary care | 4 month follow up (FU), 12 month FU
  Assessed with a Medical Report Form completed by the health care provider. "Engagement in HIV care" is operationalized as 3 visits a year (two of them at least 90 days apart) and < 2 missed visits/year

CONTACTS AND LOCATIONS:
Locations (1):
- New York University Silver School of Social Work, New York, New York, United States

REFERENCES:
- [Derived] Strayhorn JC, Cleland CM, Vanness DJ, Wilton L, Gwadz M, Collins LM. Using decision analysis for intervention value efficiency to select optimized interventions in the multiphase optimization strategy. Health Psychol. 2024 Feb;43(2):89-100. doi: 10.1037/hea0001318. Epub 2023 Aug 3. PMID 37535575
- [Derived] Gwadz MV, Collins LM, Cleland CM, Leonard NR, Wilton L, Gandhi M, Scott Braithwaite R, Perlman DC, Kutnick A, Ritchie AS. Using the multiphase optimization strategy (MOST) to optimize an HIV care continuum intervention for vulnerable populations: a study protocol. BMC Public Health. 2017 May 4;17(1):383. doi: 10.1186/s12889-017-4279-7. PMID 28472928

DOCUMENTS (1):
  • Informed Consent Form (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT02801747/ICF_000.pdf